CLINICAL TRIAL: NCT00064753
Title: Folic Acid for Vascular Outcome Reduction In Transplantation (FAVORIT)
Acronym: FAVORIT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Office of Dietary Supplements (ODS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FAVORIT dk61700 IND; U01DK061700 (NIH)
Record Dates: First submitted 2003-07-11; First posted 2003-07-15 (Estimated); Results first posted 2015-11-26 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2015-10

CONDITIONS: Chronic Kidney Disease; Cardiovascular Disease; Death
Keywords: homocysteine; multi-vitamin; cardiovascular disease; renal transplant recipients
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases; Death | interventions — Geritol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- High Dose Multivitamin (Experimental): Multivitamin with increased folic acid, vitamin B6 and vitamin B12
  Interventions: Drug: High Dose Multivitamin
- Low Dose Multivitamin (Active Comparator): Multivitamin devoid of folic acid and with estimated average requirement amounts of vitamin B6 and vitamin B12
  Interventions: Device: Low Dose Multivitamin

INTERVENTIONS:
Drug: High Dose Multivitamin — Vitamin B6 (Pyridoxine HCl): 50 mg Folic acid: 5.0 mg Vitamin B12: 1.0 mg Vitamin B1 (Thiamine HNO3): 1.5 mg Vitamin B2 (Riboflavin): 1.5 mg Vitamin C (Ascorbic Acid): 60 mg d-Biotin: 300 mcg Niacinamide: 20 mg Pantothenic Acid Calcium Pantothenate): 10 mg
  Other Names: multivitamin
  Arms: High Dose Multivitamin
Device: Low Dose Multivitamin — Vitamin B6 (Pyridoxine HCl): 1.4 mg Folic acid: 0.0 mg Vitamin B12: 2.0 mcg Vitamin B1 (Thiamine HNO3): 1.5 mg Vitamin B2 (Riboflavin): 1.5 mg Vitamin C (Ascorbic Acid): 60 mg d-Biotin: 300 mcg Niacinamide: 20 mg Pantothenic Acid Calcium Pantothenate): 10 mg
  Other Names: multivitamin
  Arms: Low Dose Multivitamin

SUMMARY:
The purpose of this randomized clinical trial is to determine if lowering homocysteine levels in renal transplant recipients with a multivitamin will reduce the occurrence of cardiovascular disease outcomes.

DETAILED DESCRIPTION:
The hypothesis of the trial is as follows: Treatment with a high dose combination of folic acid, vitamin B6, and vitamin B12 will reduce the rate of pooled arteriosclerotic cardiovascular disease outcomes (i.e., pooled occurrence of non-fatal and fatal arteriosclerotic outcomes, including coronary heart, cerebrovascular, and peripheral vascular disease events) relative to treatment with an identical multivitamin containing no folic acid, and Estimated Average Requirement amounts of vitamin B6, vitamin B12, among chronic, stable renal transplant recipients

ELIGIBILITY:
Inclusion Criteria:

* 35 - 75 years old
* Had kidney transplant at least 6 months
* Calculated Creatinine Clearance must be 25 mL/min or greater
* Must be willing to stop supplements (B6, B12, folic acid) for 4-6 weeks prior to visit

Exclusion Criteria:

* If pregnant or lactating
* If of child bearing potential and not on birth control
* If any of the following will limit life expectancy to less than 2 yrs:

  * Cancer
  * Congestive heart failure (CHF) (end stage)
  * Liver disease (end stage)
  * Severe pulmonary disease
  * Progressive HIV
  * Any other chronic wasting illness
* If patient had myocardial infarction (MI), stroke, lower extremity amputation above ankle or percutaneous revascularization procedure (coronary, cerebrovascular, lower extremity) in past 2months
* If patient had coronary artery bypass graft (CABG) or abdominal aortic aneurysm (AAA) in past 5 months
* If patient has conditions that prevent reliable study participation e.g., depression, alcohol or drug abuse, other cardiovascular disease (CVD) studies
* If patient has had multi-organ transplant, except kidney/pancreas

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4110 (Actual)
Dates: Start 2002-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Levey, M.D., Study Director — Tufts Medical Center; Myra A Carpenter, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (30):
- United States (27):
  - University of Alabama at Birmingham School of Medicine, Birmingham, Alabama
  - Banner Good Samaritan Transplant, Phoenix, Arizona
  - Cedars-Sinai Health System/Center for Kidney Diseases and Transplantation, Los Angeles, California
  - University of California at Los Angeles, Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - Northwestern University, Chicago, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Maine Medical Center, Portland, Maine
  - University of Maryland Medical Center, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Faireview University Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Albany Medical Center, Albany, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - The Ohio State University Medical Center, Columbus, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Drexel University, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Wisconsin at Madison, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Universidade Federal de Sao Paulo, São Paulo, São Paulo, Brazil
- Canada (2):
  - London Health Sciences Center, London, Ontario
  - Toronto General Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data and samples are available at the NIDDK Central repository
Supporting Information: Study Protocol, SAP, CSR
Time Frame: December 2013
URL: https://www.niddkrepository.org/studies/favorit/?query=favorit

REFERENCES:
- [Background] Weiner DE, Carpenter MA, Levey AS, Ivanova A, Cole EH, Hunsicker L, Kasiske BL, Kim SJ, Kusek JW, Bostom AG. Kidney function and risk of cardiovascular disease and mortality in kidney transplant recipients: the FAVORIT trial. Am J Transplant. 2012 Sep;12(9):2437-45. doi: 10.1111/j.1600-6143.2012.04101.x. Epub 2012 May 17. PMID 22594581
- [Background] Troen AM, Scott TM, D'Anci KE, Moorthy D, Dobson B, Rogers G, Weiner DE, Levey AS, Dallal GE, Jacques PF, Selhub J, Rosenberg IH; FACT Study Investigators. Cognitive dysfunction and depression in adult kidney transplant recipients: baseline findings from the FAVORIT Ancillary Cognitive Trial (FACT). J Ren Nutr. 2012 Mar;22(2):268-276.e3. doi: 10.1053/j.jrn.2011.07.009. Epub 2011 Dec 6. PMID 22153382
- [Background] Carpenter MA, Weir MR, Adey DB, House AA, Bostom AG, Kusek JW. Inadequacy of cardiovascular risk factor management in chronic kidney transplantation - evidence from the FAVORIT study. Clin Transplant. 2012 Jul-Aug;26(4):E438-46. doi: 10.1111/j.1399-0012.2012.01676.x. Epub 2012 Jul 9. PMID 22775763
- [Background] Bostom AG, Carpenter MA, Kusek JW, Hunsicker LG, Pfeffer MA, Levey AS, Jacques PF, McKenney J; FAVORIT Investigators. Rationale and design of the Folic Acid for Vascular Outcome Reduction In Transplantation (FAVORIT) trial. Am Heart J. 2006 Sep;152(3):448.e1-7. doi: 10.1016/j.ahj.2006.03.004. PMID 16923411
- [Background] Weir MR, Gravens-Muller L, Costa N, Ivanova A, Manitpisitkul W, Bostom AG, Diamantidis CJ; FAVORIT Study Investigators. Safety events in kidney transplant recipients: results from the folic Acid for vascular outcome reduction in transplant trial. Transplantation. 2015 May;99(5):1003-8. doi: 10.1097/TP.0000000000000454. PMID 25393158
- [Background] Carpenter MA, John A, Weir MR, Smith SR, Hunsicker L, Kasiske BL, Kusek JW, Bostom A, Ivanova A, Levey AS, Solomon S, Pesavento T, Weiner DE. BP, cardiovascular disease, and death in the Folic Acid for Vascular Outcome Reduction in Transplantation trial. J Am Soc Nephrol. 2014 Jul;25(7):1554-62. doi: 10.1681/ASN.2013040435. Epub 2014 Mar 13. PMID 24627349
- [Result] Bostom AG, Carpenter MA, Hunsicker L, Jacques PF, Kusek JW, Levey AS, McKenney JL, Mercier RY, Pfeffer MA, Selhub J; FAVORIT Study Investigators. Baseline characteristics of participants in the Folic Acid for Vascular Outcome Reduction in Transplantation (FAVORIT) Trial. Am J Kidney Dis. 2009 Jan;53(1):121-8. doi: 10.1053/j.ajkd.2008.08.010. Epub 2008 Nov 20. PMID 19022547
- [Result] Bostom AG, Carpenter MA, Kusek JW, Levey AS, Hunsicker L, Pfeffer MA, Selhub J, Jacques PF, Cole E, Gravens-Mueller L, House AA, Kew C, McKenney JL, Pacheco-Silva A, Pesavento T, Pirsch J, Smith S, Solomon S, Weir M. Homocysteine-lowering and cardiovascular disease outcomes in kidney transplant recipients: primary results from the Folic Acid for Vascular Outcome Reduction in Transplantation trial. Circulation. 2011 Apr 26;123(16):1763-70. doi: 10.1161/CIRCULATIONAHA.110.000588. Epub 2011 Apr 11. PMID 21482964
- [Derived] Kang AW, Garber CE, Eaton CB, Risica PM, Bostom AG. Physical Activity and Cardiovascular Risk among Kidney Transplant Patients. Med Sci Sports Exerc. 2019 Jun;51(6):1154-1161. doi: 10.1249/MSS.0000000000001886. PMID 30629045
- [Derived] Weinrauch LA, Claggett B, Liu J, Finn PV, Weir MR, Weiner DE, D'Elia JA. Smoking and outcomes in kidney transplant recipients: a post hoc survival analysis of the FAVORIT trial. Int J Nephrol Renovasc Dis. 2018 Apr 27;11:155-164. doi: 10.2147/IJNRD.S161001. eCollection 2018. PMID 29760559
- [Derived] Weinrauch LA, D'Elia JA, Weir MR, Bunnapradist S, Finn PV, Liu J, Claggett B, Monaco AP. Infection and Malignancy Outweigh Cardiovascular Mortality in Kidney Transplant Recipients: Post Hoc Analysis of the FAVORIT Trial. Am J Med. 2018 Feb;131(2):165-172. doi: 10.1016/j.amjmed.2017.08.038. Epub 2017 Sep 21. PMID 28943384

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial enrolled 4110 participants from August 2002 through January 2007 at 20 clinical sites in the US, Canada, and Brazil.
Groups:
- Low Dose Multivitamin: Multivitamin devoid of folic acid and with estimated average requirement (EAR) amounts of vitamin B6 and vitamin B12
  Low Dose Multivitamin: Vitamin B6 (Pyridoxine HCl): 1.4 mg Folic acid: 0.0 mg Vitamin B12: 2.0 mcg Vitamin B1 (Thiamine HNO3): 1.5 mg Vitamin B2 (Riboflavin): 1.5 mg Vitamin C (Ascorbic Acid): 60 mg d-Biotin: 300 mcg Niacinamide: 20 mg Pantothenic Acid Calcium Pantothenate): 10 mg
Period: Overall Study
Arm/Group | High Dose Multivitamin | Low Dose Multivitamin
Started | 2056 | 2054
Completed | 1382 | 1406
Not Completed | 674 | 648
Not completed — Death | 251 | 242
Not completed — Withdrawal by Subject | 198 | 171
Not completed — Lost to Follow-up | 225 | 235

BASELINE CHARACTERISTICS:
Population: 7273 patients were screened, of whom 2056 and 2054 were randomized to high-dose and low-dose multivitamins, respectively; 34% did not meet eligibility cutpoints for tHey and Cer, and 9% were not enrolled for other reasons. Baseline characteristics were well balanced between treatment groups overall and within country.
Groups:
- Low Dose Multivitamin: Multivitamin devoid of folic acid and with EAR amounts of vitamin B6 and vitamin B12
  Low Dose Multivitamin: Vitamin B6 (Pyridoxine HCl): 1.4 mg Folic acid: 0.0 mg Vitamin B12: 2.0 mcg Vitamin B1 (Thiamine HNO3): 1.5 mg Vitamin B2 (Riboflavin): 1.5 mg Vitamin C (Ascorbic Acid): 60 mg d-Biotin: 300 mcg Niacinamide: 20 mg Pantothenic Acid Calcium Pantothenate): 10 mg
- Total: Total of all reporting groups
Arm/Group | High Dose Multivitamin | Low Dose Multivitamin | Total
Number analyzed (Participants) | 2056 | 2054 | 4110
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (9.4) | 52 (9.5) | 52 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 767 | 761 | 1528
  Male | 1289 | 1293 | 2582
Region of Enrollment [Number; unit: participants]
  Canada | 249 | 249 | 498
  United States | 1500 | 1500 | 3000
  Brazil | 307 | 305 | 612
Graft vintage [Mean (Standard Deviation); unit: years] | 6 (5.1) | 5 (5.0) | 5 (5.0)
History of CVD [Number; unit: participants]
  History of CVD | 406 | 414 | 820
  No History of CVD | 1650 | 1640 | 3290
History of diabetes mellitus [Number; unit: participants]
  History of diabetes mellitus | 813 | 850 | 1663
  No history of diabetes mellitus | 1243 | 1204 | 2447
Prevalent hypertension [Number; unit: participants]
  Prevalent hypertension | 1879 | 1899 | 3778
  Non-prevalent hypertension | 177 | 155 | 332
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 29 (6.2) | 29 (6.3) | 29 (6.2)
Current smoker [Number; unit: participants]
  Current smoker | 230 | 221 | 451
  Not current smoker | 1826 | 1833 | 3659
Total cholesterol [Mean (Standard Deviation); unit: mmol/L] | 4.8 (1.2) | 4.8 (1.1) | 4.8 (1.1)
High-density lipoprotein cholesterol [Mean (Standard Deviation); unit: mmol/L] | 1.2 (0.4) | 1.2 (0.4) | 1.2 (0.4)
Calculated or direct low-density lipoprotein cholesterol [Mean (Standard Deviation); unit: mmol/L] | 2.6 (0.9) | 2.6 (0.9) | 2.6 (0.9)
Triglycerides levels [Mean (Standard Deviation); unit: mmol/L] | 2.3 (2.5) | 2.2 (1.6) | 2.2 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Recurrent or de Novo Arteriosclerotic Cardiovascular Disease (CVD) Defined as the Occurrence of Non-fatal or Fatal Arteriosclerotic Outcomes Including Coronary Heart, Cerebrovascular, and Peripheral Vascular Disease Events
Time Frame: Up to 6 years (mean 4 years)
Population: Censored at 3 months after return to dialysis
Measure: Number; unit: participants
Arm/Group | High Dose Multivitamin | Low Dose Multivitamin
Number analyzed (Participants) | 2029 | 2029
participants | 269 | 278
Statistical Analysis 1: Comparison: High Dose Multivitamin vs Low Dose Multivitamin; Test type: Superiority or Other; p = 0.93, Regression, Cox — P was calculated with stratified proportional hazards models stratified by country; Cox Proportional Hazard = 0.99, 95% CI 2-sided [0.84 to 1.17]

2. Secondary Outcome: Renal Graft Failure
Time Frame: Up to 6 years (mean 4 years)
Population: Intention-to-treat
Measure: Number; unit: participants
Arm/Group | High Dose Multivitamin | Low Dose Multivitamin
Number analyzed (Participants) | 2029 | 2029
participants | 181 | 162
Statistical Analysis 1: Comparison: High Dose Multivitamin vs Low Dose Multivitamin; Test type: Superiority or Other; p = 0.19, Regression, Cox — P was calculated with stratified proportional hazards models stratified by country; Cox Proportional Hazard = 1.15, 95% CI 2-sided [0.93 to 1.43]

3. Secondary Outcome: Mortality (All-cause)
Description: censored at 3 months after return to dialysis
Time Frame: Up to 6 years (mean 4 years)
Measure: Number; unit: participants
Arm/Group | High Dose Multivitamin | Low Dose Multivitamin
Number analyzed (Participants) | 2054 | 2049
participants | 217 | 214
Statistical Analysis 1: Comparison: High Dose Multivitamin vs Low Dose Multivitamin; Test type: Superiority or Other; p = 0.67, Regression, Cox — P was calculated with stratified proportional hazards models stratified by country; Cox Proportional Hazard = 1.04, 95% CI 2-sided [0.86 to 1.26]

4. Secondary Outcome: Fatal/Non-fatal Myocardial Infarction (MI)
Description: censored at 3 months after return to dialysis
Time Frame: Up to 6 years (mean 4 years)
Measure: Number; unit: participants
Arm/Group | High Dose Multivitamin | Low Dose Multivitamin
Number analyzed (Participants) | 2056 | 2054
participants | 90 | 86
Statistical Analysis 1: Comparison: High Dose Multivitamin vs Low Dose Multivitamin; Test type: Superiority or Other; p = 0.61, Regression, Cox — P was calculated with stratified proportional hazards models stratified by country; Cox Proportional Hazard = 1.08, 95% CI 2-sided [0.80 to 1.45]

5. Secondary Outcome: Fatal/Non-fatal Stroke
Description: censored at 3 months after return to dialysis
Time Frame: Up to 6 years (mean 4 years)
Measure: Number; unit: participants
Arm/Group | High Dose Multivitamin | Low Dose Multivitamin
Number analyzed (Participants) | 2056 | 2054
participants | 35 | 32
Statistical Analysis 1: Comparison: High Dose Multivitamin vs Low Dose Multivitamin; Test type: Superiority or Other; p = 0.64, Regression, Cox — P was calculated with stratified proportional hazards models stratified by country; Cox Proportional Hazard = 1.12, 95% CI 2-sided [0.69 to 1.81]

6. Secondary Outcome: Resuscitated Sudden Death (RSD)
Description: censored at 3 months after return to dialysis
Time Frame: Up to 6 years (mean 4 years)
Measure: Number; unit: participants
Arm/Group | High Dose Multivitamin | Low Dose Multivitamin
Number analyzed (Participants) | 2056 | 2054
participants | 7 | 9
Statistical Analysis 1: Comparison: High Dose Multivitamin vs Low Dose Multivitamin; Test type: Superiority or Other; p = 0.66, Regression, Cox — P was calculated with stratified proportional hazards models stratified by country; Cox Proportional Hazard = 0.80, 95% CI 2-sided [0.30 to 2.15]

7. Secondary Outcome: CVD Death
Description: censored at 3 months after return to dialysis
Time Frame: Up to 6 years (mean 4 years)
Population: P was calculated with stratified proportional hazards models stratified by country
Measure: Number; unit: participants
Arm/Group | High Dose Multivitamin | Low Dose Multivitamin
Number analyzed (Participants) | 2056 | 2054
participants | 75 | 91
Statistical Analysis 1: Comparison: High Dose Multivitamin vs Low Dose Multivitamin; Test type: Superiority or Other; p = 0.28, Regression, Cox; Cox Proportional Hazard = 0.84, 95% CI 2-sided [0.62 to 1.15]

8. Secondary Outcome: Coronary Artery Revascularization
Description: censored at 3 months after return to dialysis
Time Frame: Up to 6 years (mean 4 years)
Measure: Number; unit: participants
Arm/Group | High Dose Multivitamin | Low Dose Multivitamin
Number analyzed (Participants) | 2056 | 2054
participants | 111 | 120
Statistical Analysis 1: Comparison: High Dose Multivitamin vs Low Dose Multivitamin; Test type: Superiority or Other; p = 0.70, Regression, Cox; P was calculated with stratified proportional hazards models stratified by country; Cox Proportional Hazard = 0.95, 95% CI 2-sided [0.73 to 1.23]

9. Secondary Outcome: Lower Extremity Peripheral Arterial Disease (PAD)
Description: censored at 3 months after return to dialysis
Time Frame: Up to 6 years (mean 4 years)
Measure: Number; unit: participants
Arm/Group | High Dose Multivitamin | Low Dose Multivitamin
Number analyzed (Participants) | 2056 | 2054
participants | 59 | 53
Statistical Analysis 1: Comparison: High Dose Multivitamin vs Low Dose Multivitamin; Test type: Superiority or Other; p = 0.49, Regression, Cox; P was calculated with stratified proportional hazards models stratified by country; Cox Proportional Hazard = 1.14, 95% CI 2-sided [0.79 to 1.65]

10. Secondary Outcome: Carotid Endarterectomy or Angioplasty
Description: censored at 3 months after return to dialysis
Time Frame: Up to 6 years (mean 4 years)
Measure: Number; unit: participants
Arm/Group | High Dose Multivitamin | Low Dose Multivitamin
Number analyzed (Participants) | 2056 | 2054
participants | 10 | 9
Statistical Analysis 1: Comparison: High Dose Multivitamin vs Low Dose Multivitamin; Test type: Superiority or Other; p = 0.78, Regression, Cox; P was calculated with stratified proportional hazards models stratified by country; Cox Proportional Hazard = 1.14, 95% CI 2-sided [0.46 to 2.80]

11. Secondary Outcome: Abdominal Aortic Aneurysm Repair
Description: censored at 3 months after return to dialysis
Time Frame: Up to 6 years (mean 4 years)
Measure: Number; unit: participants
Arm/Group | High Dose Multivitamin | Low Dose Multivitamin
Number analyzed (Participants) | 2056 | 2054
participants | 3 | 5
Statistical Analysis 1: Comparison: High Dose Multivitamin vs Low Dose Multivitamin; Test type: Superiority or Other; p = 0.50, Regression, Cox; P was calculated with stratified proportional hazards models stratified by country; Cox Proportional Hazard = 0.61, 95% CI 2-sided [0.15 to 2.57]

12. Secondary Outcome: Renal Artery Revascularization
Description: censored at 3 months after return to dialysis
Time Frame: Up to 6 years (mean 4 years)
Measure: Number; unit: participants
Arm/Group | High Dose Multivitamin | Low Dose Multivitamin
Number analyzed (Participants) | 2 | 2054
participants | 9 | 7
Statistical Analysis 1: Comparison: High Dose Multivitamin vs Low Dose Multivitamin; Test type: Superiority or Other; p = 0.60, Regression, Cox; P was calculated with stratified proportional hazards models stratified by country; Cox Proportional Hazard = 1.30, 95% CI 2-sided [0.48 to 3.50]

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | High Dose Multivitamin | Low Dose Multivitamin
Serious Adverse Events (participants affected / at risk) | 0/2056 | 0/2054
Other Adverse Events (participants affected / at risk) | 121/2056 | 114/2054
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose Multivitamin (N=2056) | Low Dose Multivitamin (N=2054)
Gastrointestinal disturbances (Gastrointestinal disorders) | 121 | 114

LIMITATIONS AND CAVEATS:
The B-vitamin pathway for reducing total homocysteine (tHcy) may not be the optimal one for reducing CVD risk. Also, the duration of follow-up may not have been sufficient to identify a lagged impact on modification of CVD risk.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No